CLINICAL TRIAL: NCT02111252
Title: An Open-label Phase 1/2 Study to Evaluate the Safety and Immunogenicity of a Single Intramuscular Injection of TAK-850 in Healthy Adult Subjects
Brief Title: A Phase 1/2 Study of a Intramuscular Injection of TAK-850 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-850/CPH-001; U1111-1153-8702 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2014-03-11; First posted 2014-04-11 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Influenza
Keywords: Drug Therapy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-850 0.5 mL (Experimental): A single dose of 0.5 mL TAK-850 (15 µg of hemagglutinin [HA] antigen per strain) is injected into the deltoid muscle.
  Interventions: Drug: TAK-850

INTERVENTIONS:
Drug: TAK-850 — TAK-850 injection

SUMMARY:
This clinical trial is a phase 1/2 study of a single intramuscular injection of TAK-850 in healthy Japanese adult participants

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and immunogenicity of a single intramuscular injection of TAK-850 for 22 days in healthy Japanese adults

ELIGIBILITY:
Inclusion Criteria:

* 1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.

  2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.

  3. The participant is a healthy Japanese adult male or female. 4. The participant is aged 20 to 49 years, inclusive, at the time of informed consent.

  5. The participant has a body mass index (BMI) between 18.5 and 25.0 kg/m2, inclusive, at the time of eligibility evaluation.

  6. If the participant is a female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

* 1. The participant has received any investigational compound within 4 months prior to the initial injection of study vaccine.

  2. The participant has been vaccinated with seasonal influenza vaccine within 6 months prior to the initial injection of study vaccine.

  3. The participant has a history of influenza infection within 6 months prior to the initial injection of study vaccine 4. The participant is a study site employee, an immediate family member of such an employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.

  5. The participant has uncontrolled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrine or other disorders, which may impact the ability of the participant to participate or potentially confound the study results.

  6. The participant has an oral temperature ≥37.5°C prior to the initial injection of study vaccine on Day 1.

  7. The participant has any medically diagnosed or suspected immune deficient condition.

  8. The participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to the initial injection of study vaccine. Such treatments include, but is not limited to, systemic or high dose inhaled corticosteroids (>800 μg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation treatment or other immunosuppressive or cytotoxic drugs.

  9. The participant has received antipyretics within 4 hours prior to the initial injection of study vaccine.

  10. The participant has a history of Guillain- Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis) or convulsions.

  11. The participant has a functional or surgical asplenia. 12. The participant has a rash, other dermatologic conditions or tattoos which may interfere with the evaluation of injection site reaction as determined by the Investigator.

  13. The participant has a history of, or is infected with the Hepatitis B Virus (HBsAgs), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).

  14. The participant has a known hypersensitivity to any component of TAK-850. 15. The participant has a history of severe allergic reactions or anaphylaxis. 16. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the initial injection of study vaccine or is unwilling to agree to abstain from alcohol and drugs throughout the study.

  17. The participant has received any blood products (e.g. blood transfusion or immunoglobulin) within 90 days prior to the initial injection of study vaccine.

  18. The participant has received a live vaccine within 4 weeks (28 days) or an inactivated vaccine within 2 weeks (14 days) prior to the initial injection of study vaccine.

  19. If female, the participant is pregnant or lactating or intending to become pregnant before signing informed consent, during, or within 1 month after participating in this study; or intending to donate ova during such time period.

  20. The participant has donated whole blood ?200 mL within 4 weeks (28 days), ≥400 mL within 12 weeks (84 days), ≥800 mL within 52 weeks (364 days), or blood components within 2 weeks (14 days) prior to the initial injection of study vaccine.

  21. The participant has abnormal (clinically significant) electrocardiogram (ECG) at the assessment prior to the initial injection of study vaccine.

  22. The participant has abnormal laboratory values that suggest a clinically significant underlying disease at the assessment prior to the initial injection of study vaccine, or the participant has the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) more than 3 times the upper limits of normal.

  23. In the opinion of the investigator or subinvestigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reason.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Sumida-ku, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 23 March 2014 to 15 April 2014.
Pre-assignment Details: Informed consent for the study was obtained from 64 subjects in total. All subjects who gave informed consent were screened for eligibility, and 55 of these subjects were enrolled.
Period: Overall Study
Arm/Group | TAK-850 0.5 mL
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population included all participants who received treatment (full analysis set: FAS).
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Height [Mean (Standard Deviation); unit: cm] | 164.8 (7.82)
Weight [Mean (Standard Deviation); unit: kg] | 58.95 (7.185)
Body Mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.66 (1.563)
Influenza Vaccination History Within 1 Year [Number; unit: Number of participants]
  Yes | 0
  No | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Adverse Events
Description: Number of participants with injection site and systemic adverse events will be tabulated in its own, and by severity and day of onset. Described if solicited adverse event term is different from the PT.
Time Frame: For 22 days
Population: The safety analysis set, comprised the volunteers who received a single dose of 0.5 mL TAK-850, was used.
Measure: Number; unit: participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
participants
  Arthralgia | 1
  Chills | 2
  Fatigue | 1
  Headache | 3
  Injection site ecchymosis (haemorrhage) | 1
  Injection site pain | 9
  Injection site tenderness (Injection site pain) | 18
  Malaise | 9
  Myalgia | 2
  Pyrexia | 1
  Sweaty (Hyperhidrosis) | 1

2. Primary Outcome: Percentage of Participants With Seroprotection Rate of Hemagglutination Inhibition [HI] Antibody Titer
Description: Seroprotection rate is measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Seroprotection Rate was defined as the percentage of participants with HI antibody titer ≥ 40 for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain).
Time Frame: Day 22
Population: The full analysis set was used.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
Percentage of participants
  A/H1N1 strain Pre-vaccination (Day 1) | 34.5 [22.237 to 48.581]
  A/H1N1 strain 21 Days Post-vaccination (Day 22) | 81.8 [69.095 to 90.921]
  A/H3N2 strain Pre-vaccination (Day 1) | 63.6 [49.563 to 76.186]
  A/H3N2 strain 21 Days Post-vaccination (Day 22) | 87.3 [75.520 to 94.726]
  B strain Pre-vaccination (Day 1) | 20.0 [10.430 to 32.973]
  B strain 21 Days Post-vaccination (Day 22) | 76.4 [62.980 to 86.772]

3. Primary Outcome: Seroconversion Rate of HI AntibodyTiter
Description: Seroconversion rate is measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Seroconversion Rate was defined as the perccentage of participants with a baseline HI antibody titer of ≥ 10 achieving a minimal 4-fold increase, or baseline HI antibody titer of < 10 achieving an HI antibody titer of ≥ 40 for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain).
Time Frame: Day 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
Percentage of participants
  A/H1N1 strain | 70.9 [57.102 to 82.370]
  A/H3N2 strain | 52.7 [38.804 to 66.347]
  B strain | 61.8 [47.726 to 74.591]

4. Primary Outcome: Geometric Mean Fold Increase in HI Antibody Titer
Description: Geometric mean fold increase in HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination, as compared to baseline.
Time Frame: Day 22
Population: The full analysis set was used.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
Fold Change
  A/H1N1 strain | 14.74 (7.412) [8.578 to 25.335]
  A/H3N2 strain | 6.71 (6.783) [3.997 to 11.252]
  B strain7.14 | 7.14 (5.123) [4.592 to 11.108]

5. Secondary Outcome: Change From Baseline in Blood Pressure
Description: For continuous variables, summary statistics of measured values and respective changes from baseline will be calculated at each evaluation time point. In addition, figures illustrating individual changes will be created. For discrete variables, shift tables (before and after vaccination) will be created.
Time Frame: Day 1 (Baseline), Day 8, Day 22
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
mmHg
  Systolic blood pressure Day 1 | -1.2 (8.37)
  Systolic blood pressure Day 8 | -2.1 (9.23)
  Systolic blood pressure Day 22 | 0.7 (10.62)
  Diastolic blood pressure Day 1 | -2.0 (6.95)
  Diastolic blood pressure Day 8 | -2.7 (6.79)
  Diastolic blood pressure Day 22 | -2.4 (7.30)

6. Secondary Outcome: Change From Baseline in Safety Electrocardiogram (ECG) Parameters
Description: The ECG data will be analyzed into 3 categories, 'normal', 'abnormal but not clinically significant' and 'abnormal clinically significant'. Using these variables, shift tables (before and after vaccination) will be created by individual participant. . The definitions for the acronyms are as follows: Within Normal Limits (WNL), Not Clinically Significant (NCS), and Clinically Significant (CS).
Time Frame: Day 1 and Day 22
Measure: Number; unit: participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
participants
  WNL at Day 1 and WNL at Day 22 | 55
  WNL ay Day 1 and Abnormal, NCS at Day 22 | 0
  WNL at Day 1 and Abnormal, CS at Day 22 | 0
  Abnormal, NCS at Day 1 and WNL at Day 22 | 0
  Abnormal, NCS at Day 1 and Abnormal NCS at Day 22 | 0
  Abnormal, NCS at Day 1 and Abnormal, CS at Day 22 | 0
  Abnormal, CS at Day WNL at Day 22 | 0
  Abnormal, CS at Day 1 and Abnormal, NCS at Day 22 | 0
  Abnormal, CS at Day 1 and Abnormal, CS at Day 22 | 0

7. Secondary Outcome: Geometric Mean Titer (GMT) of HI Antibody Titer
Description: Geometric mean titer (GMT) of HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination
Time Frame: Day 22
Population: The full analysis set was used.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
titer
  A/H1N1 strain Pre-vaccination (Day 1) | 17.86 [10.915 to 29.209]
  A/H1N1 strain 21 Days Post-vaccination (Day 22) | 263.22 [152.753 to 453.562]
  A/H3N2 strain Pre-vaccination (Day 1) | 76.07 [42.054 to 137.592]
  A/H3N2 strain 21 Days Post-vaccination (Day 22) | 510.11 [299.040 to 870.144]
  B strain Pre-vaccination (Day 1) | 8.33 [6.342 to 10.943]
  B 21 Days Post-vaccination (Day 22) | 59.49 [39.810 to 88.908]

8. Secondary Outcome: GMT of Single Radial Hemolysis (SRH) Antibody Titer
Description: GMT of single radial hemolysis (SRH) antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination.
Time Frame: Day 22
Population: The full analysis set was used.
Measure: Geometric Mean (95% Confidence Interval); unit: mm^2
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
mm^2
  A/H1N1 strain Pre-vaccination (Day 1) | 18.1601 [12.95725 to 25.45204]
  A/H1N1 strain 21 Days Post-vaccination (Day 22) | 71.0170 [56.50806 to 89.25123]
  A/H3N2 strain Pre-vaccination (Day 1) | 7.8348 [6.13169 to 10.01108]
  A/H3N2 strain 21 Days Post-vaccination (Day 22) | 30.7917 [23.81308 to 39.81552]
  B strain Pre-vaccination (Day 1) | 32.8363 [24.66069 to 43.72228]
  B strain 21 Days Post-vaccination (Day 22) | 101.3016 [96.47024 to 106.37497]

9. Secondary Outcome: Seroprotection Rate of SRH Antibody Titer
Description: Seroprotection rate is measured by SRH antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination.
Time Frame: Day 22
Population: The full analysis set was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
percentage of participants
  A/H1N1 strain Pre-vaccination (Day 1) | 50.9 [37.071 to 64.646]
  A/H1N1 strain 21 Days Post-vaccination (Day 22) | 92.7 [82.413 to 97.983]
  A/H3N2 strain Pre-vaccination (Day 1) | 16.4 [7.766 to 28.803]
  A/H3N2 strain 21 Days Post-vaccination (Day 22) | 81.8 [69.095 to 90.921]
  B strain Pre-vaccination (Day 1) | 72.7 [59.038 to 83.862]
  B strain 21 Days Post-vaccination (Day 22) | 100.0 [93.513 to 100.000]

10. Secondary Outcome: Seroconversion Rate of SRH Antibody Titer
Description: Seroconversion rate as measured by SRH antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination.
Time Frame: Day 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
percentage of participants
  A/H1N1 strain | 81.8 [69.095 to 90.921]
  A/H3N2 strain | 74.5 [60.997 to 85.330]
  B strain | 78.2 [64.990 to 88.186]

11. Secondary Outcome: Geometric Mean Fold Increase in SRH Antibody Titer
Description: Geometric mean fold increase in SRH antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination, as compared to baseline.
Time Frame: Day 22
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | TAK-850 0.5 mL
Number analyzed (Participants) | 55
Fold Change
  A/H1N1 strain | 3.9106 (2.98684) [2.90922 to 5.25669]
  A/H3N2 strain | 3.9301 (2.75769) [2.98750 to 5.17011]
  B strain | 3.0851 (2.82759) [2.32931 to 4.08599]

ADVERSE EVENTS:
Time Frame: From the injection of study drug until 22 days.
Description: The frequencies of all adverse reactions observed during the observation period will be tabulated by type and seriousness. Adverse events are defined as unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, regardless of relationship to the medicinal product.
Arm/Group | TAK-850 0.5 mL
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 30/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-850 0.5 mL (N=55)
Injection site pain (General disorders) | 22
Malaise (General disorders) | 9
Chills (General disorders) | 2
Injection site pruritus (General disorders) | 2
Fatigue (General disorders) | 1
Injection site haemorrhage (General disorders) | 1
Injection site warmth (General disorders) | 1
Pyrexia (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.